CLINICAL TRIAL: NCT06691477
Title: A Cut-off Value Study of N-terminal Brain Natriuretic Peptide （Chemiluminescence Method）
Acronym: NT-proBNP，HF
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CHN-199
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Acute Coronary Syndromes
Keywords: NT-proBNP; Natriuretic Peptides; Diagnosis; acute heart failure; biomarker
MeSH Terms: conditions — Heart Failure; Acute Coronary Syndrome; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Remaining serum or plasma, sample volume> 500 μl
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heart Failure Cohort
  Interventions: Other: No Interventions
- Non-Heart Failure Cohort with suspected HF syndrome
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No intervention required. Subjects accepted regular medical treatment

SUMMARY:
The aim of the study is to evaluate diagnostic performance of N-terminal Brain natriuretic Peptide (NT-proBNP) in acute heart failure among Chinese population. Further, it sought to explore the optimal cut-off point fitting Chinese patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a complex clinical syndrome characterized by dyspnea, fatigue, and fluid retention (pulmonary congestion, systemic congestion, and peripheral edema) caused by abnormal changes in the structure and/or function of the heart due to multiple causes, resulting in dysfunctional ventricular contraction and/or diastolic function [1]. Heart failure is a severe or advanced stage of various cardiac diseases, with high rates of mortality and rehospitalization [1]. The prevalence of heart failure in developed countries is 1.5%~2.0%, and the prevalence in ≥ 70-year-old population ≥ 10%[2]. According to the epidemiological survey in 2003, the prevalence of heart failure in adults aged 35~74 years in China was 0.9% [3]. In recent years, with the aging of the population, the prevalence of heart failure in China has continued to increase.

A comprehensive and accurate diagnosis is a prerequisite for effective treatment for patients with heart failure, but patients with heart failure often have multiple diseases, and the clinical symptoms of heart failure overlap with those of chronic obstructive pulmonary disease and asthma, making it difficult to make clinical differential diagnosis [1]. At present, a variety of biomarkers have been used in the clinical diagnosis of heart failure, among which brain natriuretic peptide (BNP)/aminoterminal brain natriuretic peptide precursor (NT-proBNP) is the best biomarker for diagnosing heart failure [4].

Natriuretic peptides are a class of endogenous polypeptides with natriuretic and diuretic effects. BNP is an important natriuretic peptide in the human body, which is very sensitive and specifically reflects cardiac dysfunction, and has important clinical significance [5,6]. BNP is mainly synthesized by the ventricles, and when myocardial cells are stimulated, they produce a 134-amino acid B-type natriuretic peptide precursor, followed by a 108-amino acid BNP precursor, which is cleaved by the action of an endonuclease into a 76-amino acid, non-biologically active NT-proBNP, and a 32-amino acid-containing active BNP, which are released into the bloodstream [6].

Currently, blood BNP levels have been recommended by several international authoritative societies, including the American College of Cardiology Foundation/American Heart Association (ACCF/AHA), and the European Society of Cardiology (ESC), as a diagnostic and prognostic indicator of heart failure [7-10].

NT-proBNP and BNP belong to the same natriuretic peptide family and have the same biological origin. Because NT-proBNP and BNP are equimolar releases, they have similar clinical applications in the diagnosis, treatment, monitoring, and prognosis of cardiovascular diseases [5].

BNP and NT-proBNP assays were introduced in China at the beginning of the 21st century and have been widely used in clinical practice by hospitals and physicians at all levels, and have become very useful biomarkers for the diagnosis and evaluation of cardiovascular diseases, especially heart failure [6]. The 2007 Guidelines for the Diagnosis and Treatment of Chronic Heart Failure [11], the 2010 Guidelines for the Diagnosis and Treatment of Acute Heart Failure [12], and the 2018 Chinese Guidelines for the Diagnosis and Treatment of Heart Failure [1] all recommend the use of NT-proBNP and BNP for the diagnosis and prognosis of heart failure.

According to the 2018 Chinese Guidelines for the Diagnosis and Treatment of Heart Failure [1] and the ICON study [13], the cut-off values of NT-proBNP in China are as follows:

* Acute heart failure (AHF) is usually excluded with NT-proBNP < 300 ng/L;
* NT-proBNP < 125 ng/L generally excludes chronic heart failure (CHF), but its sensitivity and specificity are lower than those of AHF; • In diagnosing AHF, NT-proBNP levels should be stratified according to age and renal function: NT-proBNP levels > 450 ng/L in patients under 50 years of age, > 900 ng/L over 50 years, and > 1800 ng/L over 75 years, renal insufficiency (glomerular filtration rate < 60 mL/min) should be > 1200 ng/L.

The purpose of this study was to calculate the specificity and sensitivity of the N-terminal Brain Natriuretic Peptide Pre-Screening Test Kit (Chemiluminescence) in AHF and non-AHF* subjects at the cut-off values (300 ng/L, 450 ng/L, 900 ng/L, 1800 ng/L) for the above exclusion of AHF and diagnosis of AHF.

Note: Non-AHF means "having symptoms that would make the investigator suspect that they are related to this study, but the final diagnosis is not AHF".

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old to voluntarily participate in this study and sign the informed consent form.
* Subjects Remaining serum or plasma sample size > 500 ml.
* Have symptoms that would make the investigator suspect that they are related to heart failure.

Dyspneic patients presenting to 3 EDs in China were enrolled and had sufficient blood for subsequent NT-proBNP measurement.

Exclusion Criteria:

* Chronic kidney disease stage 4 or 5.
* Chronic renal dialysis.
* Participation in clinical studies that may interfere with participation in this study;
* Any behavior that would increase the subject's risk or prevent the subject from fully complying with or completing this study;
* The sample size is not enough for testing;
* Hemolysis, lipidemia or jaundice may be visible to the naked eye in the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Plan to 1060 Chinese patients presenting to emergency department with acute dyspnea in 3 hospitals, 2 of which are in Guangzhou and 1 in Beijing.
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy: Sensitivity and specificity | Baseline
  This study aims to evaluate the diagnostic performance of NT-proBNP for acute HF in patients with dyspnea in emergency department setting.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangzhou
  - Beckman Coulter, Shanghai, Shanghai Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - The Second Affiliated Hospital of Gungzhou Medical University, Guangzhou

IPD SHARING:
Plan to Share IPD: Undecided